CLINICAL TRIAL: NCT06720805
Title: Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Effects of a Multi-strain Probiotic in Pediatric Irritable Bowel Syndrome (PTB_IBS)
Brief Title: Pentabiocel in Pediatric IBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Di Nardo, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTB_IBS
Record Dates: First submitted 2024-11-12; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Irritable Bowel Syndrome (IBS); Pediatrics
Keywords: Irritable Bowel Syndrome (IBS); Bifidobacterium; Visceral hypersensitivity; microbiome; Lactobacillus; Pediatrics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pentabiocel (Experimental): Children with IBS who received probiotics once a day for 12 weeks.
  Every sachet contains:
  * Lactobacillus casei LMG 101/37P-17504 (5Å109 CFU/sachet)
  * Lactobacillus plantarum CECT 4528 (5Å109 CFU/sachet)
  * Bifidobacterium animalis subsp. lactis Bi1 LMG P- 17502 (10Å109 CFU/sachet)
  * Bifidobacterium breve Bbr8 LMG P-17501 (10Å109 CFU/sachet)
  * Bifidobacterium breve Bl10 LMG P-17500 (10Å~109 CFU/sachet)
  Interventions: Drug: Pentabiocel
- Placebo (Placebo Comparator): Children with irritative bowel sindrome who received placebo once a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentabiocel — This is a randomized, double-blind, placebo-controlled, multicenter clinical trial aimed at recruiting 56 pediatric patients with IBS.
  The activities will be divided into the following phases:
  1. Patient Enrollment Phase: eligible patients will meet the diagnostic criteria for IBS, as defined by internationally recognized guidelines. Informed consent will be obtained from the legal guardians of the participants before their inclusion in the study.
  2. Randomization: the enrolled participants will be randomly assigned to one of two groups: the probiotic group or the placebo group.
  3. Treatment Phase: a 3-month treatment phase will be conducted with a mixture of 5 strains of lactic acid bacteria and bifidobacter.
  4. Follow-up Phase: this will be followed by a 4-week follow-up phase. Clinical data will be monitored throughout the study using validated questionnaires.
  Arms: Pentabiocel
Drug: Placebo — This is a randomized, double-blind, placebo-controlled, multicenter clinical trial aimed at recruiting 56 pediatric patients with IBS.
  The activities will be divided into the following phases:
  1. Patient Enrollment Phase: eligible patients will meet the diagnostic criteria for IBS, as defined by internationally recognized guidelines. Informed consent will be obtained from the legal guardians of the participants before their inclusion in the study.
  2. Randomization: the enrolled participants will be randomly assigned to one of two groups: the probiotic group or the placebo group.
  3. Treatment Phase: a 3-month treatment phase will be conducted with a mixture of 5 strains of lactic acid bacteria and bifidobacter.
  4. Follow-up Phase: this will be followed by a 4-week follow-up phase. Clinical data will be monitored throughout the study using validated questionnaires.
  Arms: Placebo

SUMMARY:
Irritable Bowel Syndrome (IBS) is a common gastrointestinal disorder characterized by chronic abdominal pain and altered bowel habits, including diarrhea, constipation, or a combination of both. It is estimated to affect about 10-20% of the global population, with a higher prevalence among children and adolescents. The pathophysiology of IBS is multifactorial and involves alterations in the gut microbiota, visceral hypersensitivity, and abnormal gastrointestinal motility. Probiotics, defined as live microorganisms that provide health benefits when administered in adequate amounts, have emerged as a potential therapeutic option for IBS due to their ability to modulate the gut microbiota and exert anti-inflammatory and immunomodulatory effects.

Several studies have shown the beneficial effects of probiotics in adult IBS patients; however, few studies have been conducted in the pediatric population.

Thus, the investigators designed a randomized, double-blind, placebo-controlled, parallel-arm study evaluating the efficacy and safety of a 12-week probiotic treatment with a blend of 5 strains of lactic acid bacteria and bifidobacteria in pediatric patients with Irritative Bowel syndrome.

DETAILED DESCRIPTION:
The rationale for this study stems from the need to address the limited treatment options available for pediatric patients with IBS. Current management strategies mainly involve dietary modifications, symptomatic therapy, and psychological interventions. Probiotics offer a promising additional therapy that could potentially improve clinical outcomes and enhance the quality of life for affected children.

The specific probiotic strain selected for this study has shown beneficial effects on gut health and immune function in preclinical and clinical studies. However, its effectiveness in pediatric patients with IBS remains unexplored. Therefore, this study aims to fill this research gap by evaluating the effect of this probiotic strain on symptom severity, bowel habits, and quality of life in pediatric IBS patients.

The findings of this study could provide valuable insights into the potential therapeutic role of probiotics in pediatric IBS and contribute to the development of evidence-based guidelines for managing this condition. Furthermore, it could pave the way for additional research exploring the mechanisms of action and long-term effects of probiotics in this population, ultimately improving the overall health and well-being of pediatric IBS patients.

The theoretical framework for this study centers on understanding the potential therapeutic role of probiotics in pediatric IBS. IBS is a common gastrointestinal disorder characterized by chronic abdominal pain and disrupted bowel habits. Its pathophysiology is multifactorial, involving changes in the gut microbiota, visceral hypersensitivity, and abnormal gastrointestinal motility.

Probiotics, defined as live microorganisms that provide health benefits when administered in adequate amounts, have attracted attention as a potential treatment option for Irritable Bowel Syndrome (IBS). They have been shown to modulate the gut microbiota and exert anti-inflammatory and immunomodulatory effects. While previous studies demonstrated the beneficial effects of probiotics in adult IBS patients, few studies have been conducted in the pediatric population.

The primary motivation for this research lies in the limited treatment options available for pediatric IBS patients, which currently involve dietary modifications, symptomatic relief, and psychological interventions. Probiotics offer a promising additional therapy that could potentially improve clinical outcomes and enhance the quality of life for affected children.

Overall, the selection of this specific supplement formulation is supported by its previously demonstrated clinical efficacy, safety and tolerability, and its documented ability to modulate the gut microbiota.

To justify the use of a specific supplement formulation over others in this study, it is important to consider several factors:

1. The choice of Lactobacillus and Bifidobacterium strains was based on previous evidence showing their effectiveness in improving IBS symptoms in adults and celiac patients. The proposed formulation includes a blend of five specific strains selected for their documented ability to modulate the gut microbiota and reduce inflammation.
2. Preclinical and clinical studies have shown beneficial effects of this specific formulation in IBS patients and other gastrointestinal conditions. These preliminary data suggest that this formulation may be particularly effective in the context of pediatric IBS.
3. The safety and tolerability of this formulation have been assessed in prior clinical studies and found to be acceptable. It is important to use bacterial strains that are safe for pediatric patients and do not cause significant adverse effects.
4. This formulation has been associated with changes in the gut microbiota, including an increase in Bifidobacterium, which has been linked to improvements in IBS symptoms. This suggests that the formulation may have a positive impact on the gut microbiota composition in pediatric IBS patients.

The specific probiotic strain chosen for this study has shown favorable effects on gut health and immune function in preclinical and clinical investigations. However, its effectiveness in pediatric IBS patients remains unexplored. This study, therefore, aims to fill this research gap by evaluating the impact of this particular probiotic strain on symptom severity of symptoms, bowel habits, and quality of life in pediatric IBS patients.

To justify the absence of a comparison with another commercial probiotic in this pediatric IBS study, the following considerations were made:

1. This study is designed specifically to evaluate the efficacy of a particular probiotic formulation in pediatric IBS patients. Focusing on a single formulation allows for reduced variability in results and a more accurate assessment of the efficacy of this specific product.
2. Using multiple formulations could increase the risk of adverse effects or unwanted interactions, making safety monitoring more complex.

To justify the probiotic dosage, considering the age range (4-17 years) and the diverse weight range of subjects enrolled in the pediatric IBS study, the following factors were taken into account:

1. The selected dosage is considered safe and effective across all age and weight ranges included in the study. The investigators referred to existing preclinical and clinical data, as well as international guidelines and expert recommendations, to determine the optimal dosage for each age group.
2. The chosen dosage was set to minimize the risk of adverse effects or undesirable reactions, considering potential pharmacological interactions and long-term health impacts.

The results of this study could provide valuable insights into the potential therapeutic role of probiotics in pediatric IBS and contribute to evidence-based guidelines for managing this condition. Additionally, it may encourage further research to explore the mechanisms of action and long-term effects of probiotics in this population, ultimately leading to improved health and well-being for pediatric IBS patients.

OBJECTIVES

The primary goals of this study aim to provide evidence regarding the clinical efficacy, safety, and impact on the quality of life of the selected probiotic strain in pediatric IBS patients. The secondary objectives seek to deepen understanding of the mechanisms underlying the probiotic's long-term effects.

Primary Objectives:

1. Evaluate the effect of the probiotic on bowel habits in pediatric IBS patients. Hypothesis: Probiotic intervention will lead to an improvement in stool consistency, a reduction in the frequency of bowel movements, and a decrease in episodes of diarrhea or constipation compared to placebo.

   Hypotheses: the administration of the probiotic will lead to a significant reduction in abdominal pain, bloating, and altered bowel habits compared to the placebo.
2. Investigating the impact of the probiotic on quality of life in pediatric patients with IBS.

Hypothesis: Probiotic treatment will result in an improvement in the physical, psychological, and social aspects of quality of life for participants compared to placebo.

Secondary Objectives:

1. Evaluate the safety and tolerability of the probiotic intervention in pediatric IBS patients.

   Objective: Monitor and record any adverse events or side effects associated with probiotic treatment.
2. Assess the long-term effects of the probiotic intervention on IBS symptoms. Objective: Evaluate the sustainability of probiotic treatment effects over time.

STATISTICAL ANALYSIS

To evaluate the effect of the probiotic on bowel habits, stool consistency, frequency of bowel movements, and episodes of diarrhea or constipation, parametric or non-parametric tests will be used depending on the data distribution. For example, the Student's t-test (for normally distributed data) or the Mann-Whitney U test (for non-normally distributed data) will be used to compare the differences between the treatment group and the control group.

1. Probiotic Efficacy on Symptom Severity: To evaluate the efficacy of the probiotic in reducing symptom severity, such as abdominal pain and bloating, validated statistical tests such as Analysis of Variance (ANOVA) or equivalent non-parametric tests will be applied. This will allow the determination of significant differences between the probiotic-treated group and the placebo group.
2. Impact on Quality of Life: The impact of the probiotic on quality of life will be evaluated using specific questionnaires, such as the Bowel Habit Questionnaire and the Abdominal Pain Scale. The analysis will include descriptive statistics and appropriate tests (such as the t-test or the Mann-Whitney U test) to assess significant differences between the groups.
3. Safety and Tolerability: The safety and tolerability of the probiotic will be evaluated through the incidence of adverse events. Appropriate statistical methods, such as the Fisher's Exact Test or Chi-square test, will be used to compare the frequency of adverse events between the two groups.
4. Long-term Effects: To examine the persistence of effects over time, advanced statistical methods, such as regression analysis, will be used to assess the long-term impact of the probiotic treatment.
5. Population Analysis: All statistical analyses will be conducted on the pediatric population involved in the study, ensuring that the results are representative of the Irritable Bowel Syndrome (IBS) in this age group.

   * Significance Level: A significance level of p < 0.05 will be considered statistically significant for all tests. Confidence intervals (typically 95%) will be reported for primary and secondary outcomes to provide a better understanding of the precision of the estimates.
   * Intention-to-Treat (ITT) Analysis: An ITT analysis will be conducted, which includes all participants randomly assigned to a treatment group, regardless of whether they completed the study or adhered to the treatment protocol. This approach minimizes biases due to participants dropping out of the study and reflects the effectiveness of the probiotic treatment in the real-world setting.

SCIENTIFIC PUBLICATION PHASE OF RESULTS

1. CRF and PRO Questionnaires: A Case Report Form (CRF) will be completed with metadata and clinical information about the patients. Patients will be asked to complete questionnaires to assess the characteristics and severity of symptoms, as well as dietary and psychological factors.

   Subjects who do not complete the questionnaires will not be considered for analysis. Children aged 8 years and older will complete the forms on their own (with parental help if necessary), while children under 8 years old will have their forms completed using parent-proxy questionnaires.
2. Data Management and Protocol Compliance: The study will be conducted in compliance with the Declaration of Helsinki, the Good Clinical Practice (GCP) guidelines of the International Conference on Harmonisation (ICH), and local laws and regulations as recommended by the European Union.
3. Data Collection Tools and Source Document Identification: The Case Report Form (CRF) will serve as the primary data source. Source documentation will substantiate the integrity of the study data, confirm the recorded observations, and verify the existence of study participants. These data will be monitored with appropriate precautions to ensure confidentiality and compliance with applicable data protection laws and regulations. Staff members whose responsibilities require access to this personal data agree to maintain the confidentiality of the data.
4. Case Reporting Forms: The case reporting forms for this study are created by the principal investigator. Study data will be entered directly into the case report form by the investigator or study staff in an anonymous manner. The electronic file will be considered as the electronic Case Report Form (eCRF).

STUDY SETTING

This is a multicenter observational study. Patients will be identified through tertiary gastroenterology outpatient clinics (Fatebenefratelli Hospital ASST Fatebenefratelli Sacco in Milan and Sant'Andrea Hospital in Rome).

Potentially eligible patients will generally be identified through the following methods:

* During routine outpatient visits/consultations.
* By reviewing hospital records and databases.

ELIGIBILITY:
Inclusion Criteria:

. IBS diagnosis (all subtypes) according to Rome IV criteria

* 4 -17 years of age
* endoscopy examination (with bioptic samples) negative for IBD or microscopic colitis
* negative anti-transglutaminase antibodies
* capability to follow the protocol
* Signature of informed consent

Exclusion Criteria:

* Presence of chronic, chromosomal, or congenital anomalies, autoimmune diseases, metabolic diseases, or immunodeficiencies.
* Patients with concomitant conditions that may cognitively impair their understanding of study instructions and their ability to provide informed consent.
* Current use of non-steroidal anti-inflammatory drugs, corticosteroids, and mast cell stabilizers, use of topical or systemic antibiotics in the past month, continuous use of stimulant laxatives, major abdominal surgery, inflammatory bowel disease, infectious diarrhea, allergic diseases, and other organic or psychiatric disorders.
* Patients with concomitant organic gastrointestinal diseases (inflammatory bowel disease, celiac disease, cancer) or a major illness such as diabetes or uncontrolled thyroid disease.
* Patients with a history of intestinal surgery (excluding appendectomy or cholecystectomy).

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fecal Calprotectin Test | 3 months
  The primary outcome measure will be fFC dosage to compare bowel inflammation levels from baseline to the end of the treatment period.

SECONDARY OUTCOMES:
IBS Severity Scoring System (IBS-SSS) | 4 month
  The primary outcome will be the improvement in severity of clinical presentation from baseline to 4 weeks afer the end of the treatment period.
  Score interpretation: Remission < 75; Mild 75 -175; Moderate 175 - 300 ; Severe 300-500.
Bristol Stool Scale | 4 months
  A secondary outcome will be modifications of bowel habits from baseline to 4 weeks after the end of the treatment period.
  Scale interpretation: types 1 to 7. Types 1 and 2 constipation; types 3 and 4 ideal stools; types 6 and 7 diarrhea.
Gastrointestinal Symptom Rating Scale (GSRS) | 4 month
  A secondary outcome will be the improvement in the amount of GI symptoms from baseline to 4 weeks after the end of the treatment period.
  The GSRS is a disease-specific instrument of 15 items combined into 5 symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea and Constipation. 1 to 7 scale (1: absence of troublesome symptoms; 7: very troublesome symptoms).
IBS Quality of Life Questionnaire (IBS-QOL-34) | 4 month
  A secondary outcome will be the improvement in the quality of patients' lifestyle from baseline to 4 weeks after the end of the treatment period.
  IBS-QOL includes 34 items in a 5-point Likert scale with 8 subscales of dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual issues, and relations. The obtained scores range from 0 to 100 and it takes 10 min to complete. Higher scores indicate lower quality of life.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Ospedale Fatebenefratelli e Oftalmico, Milan
  - Ospedale Macedonio Melloni, Milan
  - Ospedale Sacco, Milan
  - Azienda Ospedaliera Sant'Andrea, Rome

IPD SHARING:
Plan to Share IPD: Undecided